CLINICAL TRIAL: NCT05371574
Title: Premedication With Oral Clonidine Versus Intraoperative Intravenous Tranexamic Acid in Reduction of Blood Loss During Elective Cesarean Section in Abakaliki - a Randomized Control Trial
Brief Title: Clonidine Versus Tranexamic Acid in Reduction of Blood Loss
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uwakwe Emmanuel Chijioke (Other)
Responsible Party: Sponsor-Investigator, Uwakwe Emmanuel Chijioke, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AEFUTHA/REC/VOLUME 3/2021/170
Record Dates: First submitted 2021-10-05; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: Will receive 100mg of tablet Vitamin C (placebo) and 1gram of intravenous tranexamic acid
Who Masked: Participant, Investigator
Masking Description: Be in brown envelop
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): Each participant will receive 1gram of tranexamic acid
  Interventions: Drug: clonidine group
- clonidine (Active Comparator): Each participant will receive 0.2mg of oral clonidine
  Interventions: Drug: clonidine group

INTERVENTIONS:
Drug: clonidine group — Each participant will be receive 0.2mg of oral clonidine 60 minutes before surgery and 10mls of sterile water (placebo) 10 minutes after skin incision
  Other Names: oral clonidine

SUMMARY:
Tranexamic acid is an antifibrinolytics agent that has been widely used in the reduction of blood loss at surgeries. Oral clonidine is an alpha-2 adrenergic agonist that has been used in various surgeries including Caesarean section.

DETAILED DESCRIPTION:
SUMMARY Background: Primary postpartum haemorrhage is a leading cause of maternal mortality and morbidity. Prevention of excessive blood loss at caesarean section is of utmost concern to the obstetrician. Blood sparing modalities are useful in the reduction of the amount of blood loss at the caesarean section. Tranexamic acid is an antifibrinolytics agent that has been widely used in the reduction of blood loss at surgeries. Oral clonidine is an alpha-2 adrenergic agonist that has been used in various surgeries including Caesarean section through its controlled hypotensive effect to reduce blood loss.

Objective: This study is designed to compare the effectiveness of Premedication with oral clonidine versus intravenous tranexamic acid in the reduction of blood loss during elective caesarean section in Abakaliki.

Methodology: This would be an equivalence double-blind, double-dummy randomized controlled clinical trial among parturients undergoing elective caesarean section in Abakaliki.This will involve 112 pregnant women at term for elective caesarean section. They will be randomized into two arms(56 Parturients in each arm). Group A will receive 100mg of tablet Vitamin C (placebo) and 1gram of intravenous tranexamic acid. Group B will receive 0.2mg of oral clonidine 60 minutes before surgery and 10mls of sterile water (placebo) 10 minutes after skin incision. The data obtained will be analysed using a statistical package for service solutions (Version 20, Chicago II, USA) and the Consolidated standard of reporting trials with the intention to treat will be applied. Continuous variables would be presented as mean and standard deviation (Mean +SD), while categorical variables would be presented as numbers and percentages. Relative Risk and logistic regression will be applied where necessary. A difference with a P-value of <0.05 will be taken to be statistically significant.

Results: The results will be presented in tables from where conclusions will be drawn.

Conclusion and Recommendation: This Will be drawn from the result.

Keyword Blood loss, Tranexamic acid, Clonidine, Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

- Participants for the study include consenting parturients with singleton pregnancy at 37-42 weeks gestational age,admitted for elective caesarean section.

Exclusion Criteria:

* Prior history of thromboembolism or bleeding disorder
* Renal disease
* Liver disease
* Antepartum Hemorrhage
* Intrauterine Growth restricted fetuses
* Patient refusal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-08-03 (Estimated); Study Completion 2022-08-03 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 6 months
  Estimated blood loss following Caesarean Section

SECONDARY OUTCOMES:
Bleeding tendency | 6 months
  Change in haematocrit 48 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Uwakwe DR Emmanuel Chijioke, PART 1, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria